CLINICAL TRIAL: NCT03737396
Title: Development and Validation of Pre-Anaesthesia CompuTerized Health Assessment (PATCH)
Brief Title: Pre-Anaesthesia CompuTerized Health Assessment
Acronym: PATCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Collaborators: Lee Kong Chian School of Medicine, National Technological University, Singapore (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: PATCH01/11/17
Record Dates: First submitted 2018-11-08; First posted 2018-11-09 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2019-10

CONDITIONS: Anesthesia; Computer, Attitude to
Keywords: Preanaesthesia health assessment; Computerized health assessment

STUDY DESIGN:
Intervention Model Description: Participating patients performs self-administered preanaesthesia health screening on an electronic tablet, before receiving nurse-administered health screening by nurses blinded to their electronic responses. This cross over study design aims to validate the electronic patient responses. In another phase, a randomized controlled trial design will be adopted to compare nurse processing time between patients who are assessed by self-administration of PATCH vs patients who undergo standard nurse-led health assessment interview.
Masking Description: In the validation phase of the study, patients, nurses and investigators are aware of participating patients' allocation in the cross over validation study. However, nurses would be blinded to the electronic responses of patients. In the randomized phase of the study, patient, nurses and investigators will be aware of group allocation and no blinding is involved.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electronic health screening (Active Comparator): Self-administered electronic health screening on tablet
  Interventions: Procedure: Self-administered electronic health screening
- Paper-based health screening (No Intervention): Routine-care nurse-administered, paper-based health screening

INTERVENTIONS:
Procedure: Self-administered electronic health screening — Health assessment using an electronic device
  Arms: Electronic health screening

SUMMARY:
Pre-anaesthesia assessment is an important component of preoperative care of surgical patients. With the increasing prevalence of same-day-admission and ambulatory surgery, patients no longer undergo preanaesthesia assessment as an inpatient in traditional "premed rounds". Currently, a nurse-administered paper-based health screening questionnaire is used at the Preadmission Service to identify patients who require outpatient evaluation by anaesthetists prior to elective surgery. In this study, the investigators aim to re-design and convert the current paper-based, nurse-administered health screening questionnaire into a reliable patient self-administered digital tool- Pre-Anaesthesia CompuTerized Health-assessment (PATCH). The electronic questionnaires will be validated by comparison of responses from digital self-administration against that obtained from a nurse interview structured to the same format. The investigators hypothesize that the responses obtained using PATCH will have at least 95% agreement with responses obtained in a nurse-led structured interview. Finally, the use of PATCH would be compared with standard nurse-led paper-based interview in a non-blinded, randomised controlled trial with regard to time taken for nurse processing of the patient at the clinic.

DETAILED DESCRIPTION:
Pre-anaesthesia assessment is an important component of preoperative care of surgical patients. Early engagement of medically-complex patients is critical to allow ample time for risk evaluation, discussion of anaesthetic plan and medical optimization. Timely and optimal preparation of patients before elective surgery could reduce morbidity and mortality, and day-of-surgery case cancellations. Due to the implementation of same-day-admission and ambulatory surgeries, medically complex patients would require preanaesthesia evaluation at an appropriate time interval prior to their elective surgery, in an outpatient facility. Currently, a nurse-administered, paper-based health screening questionnaire is used at the Preadmission Service to determine the need for outpatient specialized assessment by an anaesthetist prior to elective surgery. This process is labour-intensive and time-consuming for both patients and nurses.

The need for efficient and cost-saving processes are driving healthcare practice. Computer-assisted history-taking systems have been shown to assist clinicians in the accurate eliciting of information from patients. Increasing evidence supports the use of such systems to triage patients and determine the timing of specialist-led anaesthetic review. Low-risk patients could be evaluated by an anaesthetist on the day of surgery while high-risk patients could be channeled into appropriate pathways for evaluation and optimisation prior to day of elective surgery.

This study is planned to be conducted in several phases:

In the first phase, the investigators aim to re-design and convert the current paper-based, nurse-administered health screening questionnaire into a reliable patient self-administered digitized tool - Pre-Anaesthesia CompuTerized Health-assessment (PATCH). The feasibility of introducing a digital pre-anaesthesia health assessment screening tool will first be assessed by conducting two discrete anonymized surveys on healthcare providers and elective surgical patients to explore their needs, attitudes and acceptability towards having a digitized tool. Next, a new paper-based preanaesthesia health screening questionnaire will be designed after extensive literature review of published, validated preanaesthesia screening questionnaires and a focus group evaluation by clinicians of the anaesthesia department.

Using the draft self-administered paper questionnaire, a pilot study of about 100 patients would be conducted after obtaining written informed consent. Feedback would be sought through a short structured interview that focuses on patient's perception of language, relevance of content and ease of completion. Patients would then be processed, as per standard of care, through a nurse-led interview using the paper-based tool. Validity of each assessment question is determined by percentage agreement method. Percentage agreement of 95% or higher is considered as good criterion validity. Analysis would also include measurement of identical, contradictory and non-contradictory response rates.

In the second phase, the paper-based questionnaire will be converted to a digitized tool on an iOS platform and accessible via a tablet, called Pre-Aneshtesia CompuTerized Health assessment (PATCH). PATCH and its server would be developed using a JavaScript framework. Patient responses using self-administration of PATCH would be validated against the responses obtained by a nurse using the same platform. After written informed consent, participating patients (n=250) will complete the health screening questionnaires on a tablet without help, after which a nurse who is blinded to the patient's responses, would conduct the health screening using the same platform . Responses for each screening question will be compared for agreement and percentage agreement of 95% or higher will be considered good criterion validity.

In the final phase, a two-arm, non-blinded randomized trial would be conducted at the Preadmission Service after written informed consent, comparing duration of nurse assessment in patients who have completed the self-administration of preanaesthesia health assessment using a tablet vs those undergoing standard care nurse-led interview. Based on an expected difference in means of 3 minutes and standard deviation of 3.5 minutes at 80% power and a level of significance of 5%, the total sample size for power of analysis is 44. To account for drop-outs, the investigators aim to recruit 52 patients in this phase. Duration of nurse assessment ("service time") will be measured by the "1Q 1Payment" system and is defined from the moment the nurse clicks on the queue system to call for the patient, to completion of the nurse assessment.

Primary aim(s):

To convert a paper-based preanaesthesia health screening questionnaire into an electronic tool, with at least 95% concordance of responses from patients

To compare the duration of nurse assessment at the Preadmission Service in patients randomized to self-administration of digital preanaesthesia health assessment vs those undergoing standard nurse interview

Primary hypotheses:

The conversion of a paper-based preanaesthesia health screening questionnaire can be converted into an electronic tool, with at least 95% concordance of responses from patients.

Self-administration of a digital preanaesthesia health assessment tool does not prolong nurse assessment at the Preadmission Service, compared with standard care nurse interview.

As a secondary aim, the patients' perceptions and experience in using PATCH will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Listed for elective surgery requiring preanaesthesia health assessment at the Preadmission Service
* English-literate
* Able to use an iPad / tablet device
* Of any nationality

Exclusion Criteria:

* Patients who are severely ill or listed for emergency operations
* Visually impaired
* Not English-literate
* Unable or refuses to use an iPad / tablet device

Ages: 21 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2021-01-02 (Actual); Study Completion 2021-01-02 (Actual)

PRIMARY OUTCOMES:
Concordance of responses | 1 year
  % concordance between responses obtained from self-administration vs nurse administration of the questionnaires
Duration of nurse assessment at Preadmission Service | 1 year
  Duration of nurse assessment will be compared between digital and standard care patients

SECONDARY OUTCOMES:
Patient's perception and experience in using self-administered digital preanaesthesia health assessment tool | 1 year
  Patients' experience and perception of using PATCH would be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Eileen Lew, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No